CLINICAL TRIAL: NCT07366008
Title: The NorCUP Trial: Improving Prognosis and Personalized Treatment in Cancer of Unknown Primary (CUP)
Acronym: NorCUP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 869556
Record Dates: First submitted 2025-12-19; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Cancer of Unknown Primary Site
Keywords: cancer of unknown primary site; neoplasms, unknown primary
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Whole Genome Sequencing; Sequence Analysis, RNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comprehensive molecular profiling (Experimental): Tumor methylation analyses, cfDNA methylation analyses, Whole Genome Sequencing, RNA sequencing, Broad targeted NGS panel analyses
  Interventions: Genetic: Comprehensive molecular profiling

INTERVENTIONS:
Genetic: Comprehensive molecular profiling — A fresh frozen biopsy and blood plasma for cfDNA analyses is taken upon inclusion for comprehensive molecular profiling. Results are discussed at a study specific CUP molecular MDT meeting.
  Other Names: whole genome sequencing; RNA sequencing; Tumor methylation analyses; cfDNA methylation analyses; Broad targeted NGS panel

SUMMARY:
The goal of this clinical trial is to improve diagnosis and treatment strategies for patients with Cancer of Unknown Primary (CUP) by using advanced molecular profiling to identify the likely tumor origin and guide therapy.

The main questions it aims to answer are:

Can comprehensive molecular profiling help determine the origin of CUP tumors? Does identifying the tumor origin improve treatment choices and survival outcomes compared to historical data?

Participants will:

* Undergo a new biopsy to collect tumor tissue for advanced analyses.
* Provide blood samples for circulating tumor DNA (cfDNA/ctDNA) analyses.
* Provide a fecal sample for microbiome analysis.
* Have their tumor tissue analyzed using:

Methylation profiling and comprehensive gene panel testing.

* Have the results reviewed in a specialized CUP molecular MDT meeting to determine the likely tumor origin and guide treatment.
* Have their tumor tissue samples biobanked for further exploratory whole genome sequencing (WGS) and RNA sequencing.

ELIGIBILITY:
Inclusion Criteria:

* ECOG PS 0-2.
* Life expectancy minimum 3 months.
* Radiologically verified metastatic disease (CT thorax/abdomen/pelvis) with no radiological signs of primary tumor.
* Histologically verified metastatic disease of unknown primary. Morphological and immunohistochemical findings suggesting a possible, but not definitive, origo is eligible.
* Eligible histologies include adenocarcinoma, squamous cell carcinoma, poorly and undifferentiated carcinoma and undifferentiated neoplasms.
* Clinically relevant endoscopic examinations have been performed as indicated by clinical, radiological and pathological findings, without identification of a primary tumor.
* Clinically relevant supplementary radiological examinations have been performed as indicated by clinical, radiological and pathological findings, with no radiological signs of primary tumor (e.g. PET/CT, mammography/MR mammae).
* Metastatic lesion available for biopsy. Protocol deviation may be allowed if lesion is not technically available for biopsy. For patients with metastatic lesion technically available for biopsy, the patient must be deemed medically fit to undergo a metastatic biopsy, as assessed by the investigator.
* Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* Patients with any clinically significant medical or psychiatric condition which, in the opinion of the treating physician, makes it undesirable for the patient to participate in the study or which could jeopardize compliance with study requirements.
* Psychological, familial, sociological or geographical condition(s) potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Patient not able to give an informed consent or comply with study regulations as deemed by study investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2033-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients where the site of origin is identified | From enrollment to the conclusion at the CUP molecular MDT at 8 weeks
  Site of origin identified is defined as the cases where the CUP molecular MDT concludes with a likely primary site of origin
Percentage of patients where treatment choice differs from empirical CUP regimen | From conclusion at the CUP molecular MDT to the start of subsequent treatment within a timeframe of 36 months from study inclusion
  Organ specific treatment chosen over empirical CUP treatment, based on the conclusion from the CUP MDT

SECONDARY OUTCOMES:
Progression free survival | From the date of first administration of a treatment line to the date of progression or death, or censored if alive at time of analysis, with a timeframe of 36 months from study inclusion.
  The length of time from the start of treatment until disease progression or death from any cause, whichever occurs first.
Overall survival | From date of CUP diagnosis until death from any cause or censored if alive at date of analysis, within a timeframe of 36 months from study inclusion.
  Length of time from CUP diagnosis until death from any cause
Identification of tumor site using molecular profiling methods | From study enrollment to the conclusion at the CUP molecular MDT at 8 weeks
  The percentage of patients in whom the likely site of origin is identified by each molecular profiling method.
Incidence of molecular alterations and use of targeted treatment in CUP patients | From molecular profiling to initiation of targeted therapy and follow-up for survival outcomes, within a timeframe of 36 months from study inclusion.
  The frequency of molecular alterations and actionable targets in patients with CUP, and the percentage of patients receiving targeted therapy based on molecular profiling results. The impact of targeted treatment on survival will also be evaluated.
Impact of CUP molecular MDT assessement on previous clinical work-up | From enrollment until CUP mol MDT at 8 weeks
  This outcome evaluates the utility of CUP molecular MDT meetings by measuring the percentage of patients for whom additional clinical work-up or pathology analyses are recommended and the concordance between local and study pathologist conclusions.

OTHER OUTCOMES:
Fecal Microbiome Diversity and Composition in CUP Patient | From baseline stool sample collection through completion of analyses within a timeframe of 36 months from study inclusion
  Characterization of the fecal microbiome in patients with cancer of unknown primary (CUP)

CONTACTS AND LOCATIONS:
Locations (6):
- Norway (6):
  - Haukeland University Hospital, Bergen
  - Akershus University Hospital, Oslo
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of North-Norway, Tromsø
  - St Olavs Hospital, Trondheim